CLINICAL TRIAL: NCT04982991
Title: A Phase 1, Open-label, 3-treatment Period, 1-sequence, Cross-over Study of the Pharmacokinetics, Safety and Tolerability After Single Ascending Oral Doses of SAR443820 in Healthy Adult Chinese and Japanese Female and Male Participants.
Brief Title: Single Ascending Dose Study of SAR443820 in Healthy Adult Chinese and Japanese Female and Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PKM17247; 2021-001076-42 (EudraCT Number); U1111-1264-3008 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04-08

CONDITIONS: Multiple Sclerosis Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAR443820 (Experimental): Participants will receive a single sequence of 3 different doses of SAR443820 in a total of 3 treatment periods
  Interventions: Drug: RIPK1 inhibitor

INTERVENTIONS:
Drug: RIPK1 inhibitor — Capsule Oral
  Other Names: SAR443820

SUMMARY:
Primary Objective:

To assess the pharmacokinetic parameters of SAR443820 after ascending single oral doses in healthy East Asian (Chinese and Japanese) adult participants.

Secondary Objective:

To assess the tolerability and safety of SAR443820 after ascending single oral doses in healthy East Asian (Chinese and Japanese) adult participants

DETAILED DESCRIPTION:
The duration of the study for a participant will be up to approximately 7 weeks and include:

* Screening period: up to 4 weeks (Day -28 to Day -2).
* Institutionalization period at each period of treatment: 4 days (Day -1 to Day 3, single SAR443820 administration on Day 1).
* Wash-out period: at least 5 days between each dosing.
* End-of-study visit: Period 3/ Day 6±1 day.

ELIGIBILITY:
Inclusion Criteria:

East Asian (Chinese and Japanese) male and/or female participant must be 20 to 55 years of age inclusive, at the time of signing the informed consent.

Chinese or Japanese ethnicity, according to the following criteria:

Chinese; born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China.

Japanese; born in Japan or ethnic Japanese born outside of Japan, and a descendent of 4 ethnic Japanese grandparents who were all born in Japan.

Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG.

Body weight within 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, and body mass index (BMI) within the range 18.0 and 30.0 kg/m2, inclusive.

Exclusion Criteria:

Medical history of any seizure.

Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, any live attenuated vaccine given within 3 months or any non-live vaccine given within 2 weeks before inclusion, and any biologics (antibody or its derivatives) given within 4 months before inclusion.

Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test.

Current psychiatric disorder, suicidal ideation in the previous 6 months (as assessed by the Columbia-Suicide Severity Rating Scale [C-SSRS]), or a lifetime suicide attempt. A "yes" response to questions 4 or 5 on the Suicidal Ideation section, or a score of 4 or 5 on the Intensity of Ideation section of the baseline/screening version of the C-SSRS at screening, or on the Since Last Visit version of the C-SSRS at baseline.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetic (PK) parameter: Cmax | Up to day 3
  Maximum plasma concentration
Assessment of pharmacokinetic (PK) parameter: AUClast | Up to day 3
  Area under the plasma concentration versus time curve from time zero to the real time last
Assessment of pharmacokinetic (PK) parameter: AUC | Up to day 3
  Area under the plasma concentration versus time curve

SECONDARY OUTCOMES:
Assessment of adverse events (AEs) | Up to day 21
  Number of participants with Adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site Number :8260001, Harrow, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org